CLINICAL TRIAL: NCT04356768
Title: Routine Histological Analysis of Sacrococcygeal Pilonidal Sinus Specimens, Retrospective Analysis of 1971 Resections.
Brief Title: Histological Analysis of Sacrococcygeal Pilonidal Sinus Specimens
Status: Completed | Type: Observational
Sponsor: Dr. Ersin Arslan Education and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Uylas, Specialist, Dr. Ersin Arslan Education and Training Hospital
Other Study IDs: 17042020
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pathology
Keywords: Pilonidal sinus; carcinoma; pathology; squamous cell carcinoma; phenol
MeSH Terms: conditions — Pilonidal Sinus; Carcinoma; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Minimally invasive techniques have been widely used routinely and reliably in the treatment of pilonidal sinus. In some of these methods, the cavity of sinus remains in the patient; this condition caused us to question the necessity of pathological examination. Except for prolonged duration of disease, elderly age, macroscopic suspicion, and recurrence; We think that routine pathological examination of the pilonidal sinus is unnecessary.

DETAILED DESCRIPTION:
Pilonidal sinus is a benign disease. In the histopathological examination of pilonidal sinus specimens, malignancy can be detected rarely. Minimally invasive techniques have been widely used routinely and reliably in the treatment of pilonidal sinus. In some of these methods, the cavity of sinus remains in the patient; this condition caused us to question the necessity of pathological examination. The investigators aimed to discuss the pathological findings of patients who were operated for pilonidal sinus in our clinic in light of the literature. The fact that the rate of malignancy in the literature does not show parallelism with minimally invasive procedures that pathology samples are not taken and whose applications are increasing supports this prediction. Except for prolonged duration of disease, elderly age, macroscopic suspicion, and recurrence; the investigators think that routine pathological examination of the pilonidal sinus is unnecessary.

ELIGIBILITY:
Inclusion Criteria:

* sacrococcygeal pilonidal sinus

Exclusion Criteria:

* non-sacrococcygeal pilonidal sinus
* minimally invasive treatment without histopathological examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were operated on for pilonidal sinus between January 2016 and March 2020 at our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1971 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Incidental cancer | 2 or 3 week
  Routine Histological Analysis of Sacrococcygeal Pilonidal Sinus Specimens

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Uylas, Specialist, Principal Investigator — Dr. Ersin Arslan Training and Resource Hospital
Locations (1):
- Dr. Ersin Arslan Training and Resource Hospital, Gaziantep, Turkey (Türkiye)